CLINICAL TRIAL: NCT03205020
Title: Maternal Serum Amyloid A Levels in Pregnancies Complicated With Preterm Labour.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: mona nematallah (Other)
Responsible Party: Sponsor-Investigator, mona nematallah, physician, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: amyloid a
Record Dates: First submitted 2017-06-13; First posted 2017-07-02 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with preterm labor
  Interventions: Diagnostic Test: serum amyloid a test
- women delivered at full term
  Interventions: Diagnostic Test: serum amyloid a test

INTERVENTIONS:
Diagnostic Test: serum amyloid a test — * Women who are diagnosed with preterm labor (28-36 weeks) will be enrolled in this study. Serum samples will be collected from all women before any intervention. All women will be sampled once at the time of admission.
  * Venous blood sample (5 c.c) will be taken from each participant for examination of serum amyloid A.
  * The collected blood will be centrifuging and serum will be stored to measure the level of amyloid A by (ELISA) technique in clinical pathology department- Ain shams University

SUMMARY:
The aim of the current study is to assess the accuracy of maternal serum amyloid A for prediction of preterm labor in women with threatened preterm labor.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, age 18 - 35.
* Gestational age: 28 - 36+6 weeks.
* Singleton pregnancy.
* No past history of any medical disorder and with no other medical complications during pregnancy
* Nonsmoker.
* Diagnosis of preterm labor is based on the American College of Obstetricians and Gynecologists Guidelines

Criteria of preterm delivery:

1. Gestational age: 28 - 36+6 weeks
2. Presence of uterine contractions (at least 4 in 20 minutes or 8 in 60 minutes)
3. cervical dilation ≥ 4 cm
4. Cervical effacement ≥ 80%.

Exclusion Criteria:

* Of any patient with the following risk factors for preterm labor:

  * Over distended uterus .
  * hemorrhage
  * Uterine anomalies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 58 pregnant women will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of Amyloid A level in women with preterm labour | 6 months
  venous sample will be taken from each participant from onset of labour, Amyloid a level will be calculated

SECONDARY OUTCOMES:
neonatal complications | 6 months
  preterm baby will be examined at neonatal intensive care unit by neonatologist.
  • Admission to Neonates intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: mona mohamed, MS, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pubmed/25118503